CLINICAL TRIAL: NCT00715143
Title: Post Approval Study: NOVATION Ceramic Articulation Hip System A Multi-Center, Open-Label Study to Evaluate the Mid and Long-Term Safety and Effectiveness of the Exactech NOVATION Ceramic Articulation Hip System
Brief Title: Post Approval Study: NOVATION Ceramic Articulation Hip System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Exactech withdrew the PMA associated with the study device due to low market utilization
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR05-005
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2015-02

CONDITIONS: Total Hip Replacement (Non-inflammatory)
Keywords: hip; replacement; ceramic; orthopaedic; joint; degenerative; non-inflammatory; osteoarthritis; avascular necrosis; congenital hip dysplasia; traumatic arthritis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Hip Dislocation, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects will be receive the Novation Ceramic on Ceramic Articulating Hip System (Other): All subjects will receive the Novation Ceramic on Ceramic Articulating Hip System.
  Interventions: Device: Novation Ceramic

INTERVENTIONS:
Device: Novation Ceramic — This treatment is the study device (which will be compared to a similar historic control device)
  Other Names: Novation

SUMMARY:
The purpose of this study is to collect and evaluate long-term safety and effectiveness data on the Exactech® NOVATION ™ Ceramic Articulation Hip System ("NOVATION ™ Ceramic AHS").

DETAILED DESCRIPTION:
The purpose of this study is to collect and evaluate long-term safety and effectiveness data on the Exactech® NOVATION ™ Ceramic Articulation Hip System ("NOVATION ™ Ceramic AHS"). Ten (10) years of follow-up data will be collected in this study. The first five (5) years of subject follow-up will involve clinical (Harris Hip Score, adverse events), radiographic, and self-assessment evaluation. The remaining five (5) years of subject follow-up will be accomplished with an outcomes questionnaire that will be completed by the subjects to evaluate the survivorship status of their hip replacement.

ELIGIBILITY:
Inclusion Criteria

1. Patient is undergoing primary hip surgery for symptomatic Non-inflammatory Degenerative Joint Disease (NIDJD). Composite diagnosis of NIDJD includes osteo/ degenerative arthritis, traumatic arthritis, congenital hip dysplasia and avascular necrosis.
2. Patient is 21 years of age or older at the time of surgery.
3. Patient is skeletally mature (tibial and femoral epiphyses are closed).
4. Patient is willing and able to return for follow-up as specified by the study protocol over a ten (10) year post-operative follow-up period; including 5 years of in-clinic visits followed by 5 years of mail-in questionnaire follow-up.
5. Patient is female and of childbearing age, for whom a negative urine pregnancy test is obtained immediately prior to surgery.
6. Patient does not meet any of the Exclusion Criteria.
7. Patient agrees to participate and sign the Informed Consent Form.

Exclusion Criteria

1. Patient will be less than 21 years old at the time of surgery.
2. Patient is skeletally immature.
3. Patient presents with inflammatory degenerative joint disease.
4. Patient has evidence of active infection, but not including asymptomatic urinary tract infection (UTI) if treated with antibiotics preoperatively.
5. Patient is female and of child bearing age and is pregnant or whose pregnancy status is unknown.
6. Patient has neurological or musculoskeletal disease that may adversely affect gait or weight bearing.
7. Patient has known presence of active metastatic or neoplastic disease (active is defined as within the past 5 years. Does not include basal cell carcinoma in cases when a subject with this diagnosis has undergone radical excision of the lesion, has pathological proof that the lesion has clean and clear peripheral and deep borders, and the location of the lesion is not near the operative hip or on the affected extremity).
8. Patient has poor bone quality (e.g., osteoporosis) where, in the investigator's opinion, there is inadequate bone to support the implant(s).
9. Patient has the presence of a previous prosthetic hip replacement device (any type, including THA, surface replacement arthroplasty, endoprosthesis, etc.) in the operative hip joint.
10. Patient is known to have presence of a highly communicable disease or diseases that may limit follow-up (e.g., immuno-compromised conditions, hepatitis, active tuberculosis, etc.).
11. Patient is a prisoner.
12. Patient is obese where obesity is defined as a Body Mass Index (BMI) greater than 35. BMI = Weight (lbs.) ÷ Height (in.)2 x 703
13. Patient has neuropathic joints.
14. Patient has known allergies to the implant materials.
15. Patient is unwilling or unable to comply with postoperative rehabilitation instructions and weight bearing limitations.
16. Patient's life expectancy is < 5 years due to chronic diseases such as cancer, congestive heart failure, etc.
17. Patient is unwilling or unable (e.g. cases of reduced mental capacity) to return for follow-up as specified by the study protocol over a ten (10) year post-operative follow-up period.
18. Patient has reduced mental capability (permanent or temporary) that would prevent following pre-surgical and post-surgical instructions.
19. Patient otherwise meets the study criteria but refuses to consent in writing to participate in the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-06; Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Radiographic evaluation of radiolucency | Immediately post operation, 6 weeks, 6 months, annually 1-5 years
  Radiographic analysis
Survivorship of device components | Immediately post operation, 6 weeks, 6 months, annually 1-5 years
  Device Survivorship
Harris Hip Score | Immediately post operation, 6 weeks, 6 months, annually 1-5 years
  Physician assessed outcome

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Shrock Orthopedic Research, Fort Lauderdale, Florida
  - Resurgens Orthopaedics, Cumming, Georgia
  - Fallon Clinic, Worcester, Massachusetts
  - Tulsa Bone & Joint Associates, Tulsa, Oklahoma
  - Hampton Roads Orthopaedics & Sports Medicine, Newport News, Virginia